CLINICAL TRIAL: NCT00671944
Title: Long-term Impact of Protein on Calcium Kinetics
Brief Title: Long-term Nutritional Intervention Study to Determine How Protein Affects Calcium Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Karl Insogna, MD, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304025163
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Osteoporosis
Keywords: protein; calcium; parathyroid hormone; bone markers; calcium kinetics; absorption
MeSH Terms: conditions — Osteoporosis | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Low protein diet
  Interventions: Other: Low protein diet

INTERVENTIONS:
Other: Low protein diet — Low protein diet for 6.5 weeks

SUMMARY:
Osteoporosis is a major health problem in men and women in this country and the incidence of this disease is rising. We think that environmental factors such as nutrition may play a role in the increasing prevalence of osteoporosis. In particular, we think that a diet that is too low in protein may be contributing to bone loss. The primary purpose of this study is to compare the long-term impact of a low protein diet on measures of bone and calcium metabolism.

DETAILED DESCRIPTION:
The protocol is composed of a 9.5-week study, consisting of a 3-week adjustment period followed by a 6.5-week experimental period. During the adjustment period, subjects consume a well-balanced lead-in diet designed to stabilize baseline Ca homeostasis. In the subsequent experimental period, subjects will consume the experimental diet containing 0.7 g protein/kg, 800-1200 mg phosphorus, 800 mg calcium and 2300 mg sodium. During days -6 to -1 of the adjustment diet, 5-10 and days 40-45 of the experimental period, we will measure Ca absorption and kinetics. Weekly assessments of Ca homeostasis will be done using our standard measures of calcitropic hormones, markers of bone turnover, and urine and serum minerals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Asian or Caucasian women between the ages of 20-40 years.

Exclusion Criteria:

* Diseases or medical conditions: gastrointestinal diseases, osteoporosis, diabetes, hypertension, liver disease, thyroid disorders, kidney disease, kidney stones, cancer, heart disease, eating disorders, obesity, hypogonadism , amenorrhea, oligomenorrhea, abnormal serum FSH or estradiol levels, birth control medication, or other hormone-altering medications, pregnancy.
* Lifestyle: smoking, excessive exercise (although moderate exercise is allowed), prescription medications known to influence vitamin D or calcium metabolism or gastric acid, excessive body weight change during the past 6 months, food allergies, unusual eating habits, or medically prescribed diets.
* Also excluded are prisoners and individuals who are cognitively impaired.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2003-05; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Calcium absorption and kinetics | Baseline, day 5 and week 6

SECONDARY OUTCOMES:
Serum Parathyroid hormone | baseline and weekly
Markers of bone turnover | baseline and weekly

CONTACTS AND LOCATIONS:
Overall Officials: Karl L Insogna, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Research Unit, New Haven, Connecticut, United States